CLINICAL TRIAL: NCT00217178
Title: Homocysteine Lowering and Atherosclerosis Reduction Trial (HART)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Population Health Research Institute (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HART, CIHR Grant # MCT 44159; CIHR, MCT 44159
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2004-10

CONDITIONS: Atherosclerosis; Cardiovascular Disease
Keywords: Atherosclerosis; CV Risk Factors; Homocysteine; CV disease; Cardiovascular disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Vitamin B 12

INTERVENTIONS:
Drug: Vitamins: Folic acid, B6, B12

SUMMARY:
Study Objective:

1. To evaluate whether combined therapy with folic acid 2.5 mg/day, vitamin B6 50 mg/day and vitamin B12 1000 micrograms/day vs placebo reduces the rate of atherosclerosis progression, as evaluated by quantitative B-mode carotid ultrasound (US).

DETAILED DESCRIPTION:
The HART study is designed as a substudy of the Heart Outcomes Prevention Evaluation-2 (HOPE-2)trial which evaluates the effect of combined therapy ? folic acid and vitamin B6 and B12 on clinical events. The study is designed to enrol 900 study participants randomized to homocysteine lowering therapies or placebo. Follow-up will estimate over 5 years. Study participants will undergo yearly carotid B-Mode ultrasound examinations.

ELIGIBILITY:
Inclusion Criteria:Women and Men aged ≥ 55 years at high risk for CV events with: (a) Documented (CAD): i) History of prior MI; ii) stable or unstable angina with documented multivessel CAD or strongly positive stress test; iii) Multivessel CAD and PTCA ≥ 6 months prior to randomization; iv) multivessel CABG ≥ 4 years prior to randomization; v) Multivessel CAD on angiography; (b) Documented peripheral vascular disease (PVD): i) Previous limp bypass surgery and/or previous peripheral percutaneous transluminal angioplasty and/or previous limp or foot amputation due to PVD.ii) History of intermittent claudication with ankle/arm blood pressure ratio of ≤ 0.80 or with significant arterial stenosis on angiography; (c) Documented cerebrovascular disease: i) History of previous ischemic stroke; and (d) Diabetes mellitus with ≥ 1 additional major CV risk factor(s). (2) Provision of informed consent.(3) Adequate baseline carotid US examination.

Exclusion Criteria:1. Current use of folic acid supplements > 200 mg/day. 2. Known previous adverse reactions to folic acid, Vitamin B6 or B12. 3. Planned cardiac, peripheral or cerebrovascular.

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2000-01; Study Completion 2005-10

PRIMARY OUTCOMES:
The change over time (annualized progression slope) in the mean maximum IMT (the mean maximum IMT slope) defined as the average of the maximum IMT across the 12 preselected carotid arterial segments.

SECONDARY OUTCOMES:
The change over time (annualized progression slope) in the single maximum IMT amongst any of the same preselected carotid artery segments, i.e. the hemodynamically most important lesson.

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Lonn, MD MSc FRCPC FACC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences Corp., Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Held C, Sumner G, Sheridan P, McQueen M, Smith S, Dagenais G, Yusuf S, Lonn E. Correlations between plasma homocysteine and folate concentrations and carotid atherosclerosis in high-risk individuals: baseline data from the Homocysteine and Atherosclerosis Reduction Trial (HART). Vasc Med. 2008 Nov;13(4):245-53. doi: 10.1177/1358863X08092102. PMID 18940900